CLINICAL TRIAL: NCT03601845
Title: Magnetic Resonance Elastography by Intrinsic Activation in Liver Disease and Neurovascular Imaging
Brief Title: MRE-IA in Liver Disease and Neurovascular Imaging
Acronym: MRE-IA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Centre hospitalier de l'Université de Montréal (CHUM) (Other); Réseau de bio-imagerie du Québec (RBIQ) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MEO-31-2019-7773
Record Dates: First submitted 2018-06-18; First posted 2018-07-26 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Diffuse and Focal Liver Diseases, Cerebral Function
Keywords: Magnetic resonance elastography; Intrinsic activation; Liver disease; Cerebral function
MeSH Terms: conditions — Liver Diseases | interventions — Stimuli Responsive Polymers

STUDY DESIGN:
Intervention Model Description: Additional sequences during magnetic resonance elastography by intrinsic activation with or without stimuli
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRE-IA (no stimuli) (Other): Additional sequencing only
  Interventions: Other: No stimuli
- MRE-IA with stimuli (Active Comparator): Visual stimulation while using additional sequencing
  Interventions: Other: Stimuli

INTERVENTIONS:
Other: Stimuli — Visual stimulation while using additional sequencing
  Arms: MRE-IA with stimuli
Other: No stimuli — Additional sequencing only
  Arms: MRE-IA (no stimuli)

SUMMARY:
The objective of this research project is to develop Magnetic Resonance Elastography by Intrinsic Activation (MRE-IA) imaging methods at two imaging centers (CRCHUS and CRCHUM) for use in ongoing studies in liver disease and neurovascular imaging. MRE is a developing MR imaging modality that provides detailed maps of tissue's mechanical properties, based on displacement measurements made during the propagation of low amplitude vibrations through the region of interest. MRE-IA uses the pressure pulses of the cardiac cycle to induce the vibrations needed for MRE image reconstruction.

MRE-IA has already been demonstrated based on the use of existing, clinically approved MR imaging sequences, and once this capability has been established at the two centers, initial trials will be done to demonstrate the method's potential in liver and neurovascular imaging. In the case of the liver, this pilot project funding will be used to perform MRE-IA imaging in patients with chronic liver disease and focal liver lesions. Results will be analyzed to establish the relationship between the mechanical properties mentioned above and disease stage. In the neurovascular case, imaging will be conducted under basic visual and motor stimulus conditions in healthy subjects, and results compared non-stimulus control images to determine changes in the above properties based on brain function. In addition, MRE-IA images will be compared with BOLD imaging to investigate the role of fluid conductivity in fMRI results.

DETAILED DESCRIPTION:
Unlike current MRE methods which require the application of cyclical mechanical excitations with an external driver, MRE-IA is a recently developed MRE modality that uses the naturally occurring cardiac pressure cycle to generate the displacements used for elastic property reconstruction. With no external activation, MRE-IA provides a simple pathway towards in-vivo elastography results that avoids the discomfort, poor coupling, and high attenuation often observed in MRE extrinsic vibration drivers.

Goals: The principal goal of this project is to establish Magnetic Resonance Elastography by Intrinsic Activation (MRE-IA) imaging methods at the imaging centers of the Centre de recherche du centre hospitalier universitaire de Sherbrooke (CRCHUS) and the Centre de recherche du centre hospitalier universitaire de Montréal (CRCHUM). Each imaging center will then focus on separate sub-goals: improving liver disease assessment with MRE-IA (CRCHUM) and evaluating the role of fluid conductivity and changes in elastic properties with mental tasks (CRCHUS).

Hypothesis: There are two main hypotheses underlying this project: (1) that internal activation provides an effective, robust displacement source for MRE image reconstruction that eliminates the problems of discomfort, high attenuation, artefact sensitivity, and low signal to noise associated with traditional extrinsic MRE methods; and (2) that the advanced material property maps provided by MRE-IA, such as viscoelastic damping, poroelastic effects and anisotropy, will lead to better classification and understanding of both diseased and healthy tissue states.

Methods: The image acquisition methodology for this project will be identical at both imaging centers. Intrinsic activation MRE displacement data will be obtained through the use the Q-Flow angiographic sequence available on the Philips 3T systems at both the CRCHUS and CRCHUM.

MRE-IA for diffuse and focal liver disease (CRCHUM): The objective of this study is to demonstrate the feasibility of MRE-IA imaging in the assessment of liver disease. MRE-IA will be performed in three populations (10 healthy volunteers, 25 patients with diffuse liver disease and 10 patients with focal liver lesions)

Intrinsic MRE: MRE-IA images are reconstructed from phase-contrast sequences that are currently available on MRI scanners at CHUM and CHUS. Post-processing of the images with finite element analysis (FEA) mechanical simulations allows calculation of poroviscoelasticity parameters (i.e. porosity, bulk modulus, storage modulus [G'], and loss modulus [G'']). These poroviscoelasticity parameters will be correlated with histopathological markers of disease severity (fibrosis, inflammation, fat) in patients with chronic liver disease and with the final diagnosis (type of liver lesion).

Cerebral function imaging via MRE-IA (CRCHUS): The objective of this study is to investigate the changes in mechanical properties during the performance of mental tasks and the role of inherent fluid conductivity in the BOLD imaging used in fMRI methods. Multiple imaging sessions will be performed to investigate changes to MRE-IA property maps to visual (V1) stimulation. Imaging sessions will be include either V1 (n=6) or non-stimulus (n=3) cases. Each case will include both MRE-IA and fMRI acquisitions.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years old at screening;
* Are able to comprehend and willingness to provide voluntary consent;
* Are able to have a MRI;
* Understand French or English;
* At CHUM:

  * Healthy volunteers or;
  * Have a diffuse liver disease (non alcoholic cirrhosis, hepatitis, NASH) and

    * Are scheduled for liver biopsy as part of their standard of care
    * Are scheduled for a MRI for clinical or research purpose, or;
  * Have a focal liver lesion (e.g. hemangioma, hepatocellular carcinoma, cholangiocarcinoma, and metastases) and

    * Are scheduled for clinical MRI as part of their standard of care for characterization of liver masses
* At CHUS:

  * Healthy volunteers.

Exclusion Criteria:

* Have a contra-indication for MRI (such as claustrophobia, pacemaker, metallic clips for a neurosurgical procedure);
* Are pregnant or trying to become pregnant;
* Have a weight or girth preventing them from entering the MR magnet bore;
* Are unable to understand or unwilling to provide written informed consent for this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Elasticity of brain | 1 day During scheduled brain iMRE examination
  Measure of elasticity of brain using iMRE
Viscosity of brain | 1 day During scheduled brain iMRE examination
  Measure of viscosity of brain using iMRE
Porosity of brain | 1 day During scheduled brain iMRE examination
  Measure of porosity of brain using iMRE
Elasticity of liver | 1 day During scheduled brain iMRE examination
  Measure of elasticity of liver using iMRE
Viscosity of liver | 1 day During scheduled brain iMRE examination
  Measure of viscosity of liver using iMRE
Porosity of liver | 1 day During scheduled brain iMRE examination
  Measure of porosity of liver using iMRE

SECONDARY OUTCOMES:
Correlation between measures of poroviscoelasticity parameters of liver and histopathological features | 1 day During scheduled brain iMRE examination
  Measure of correlation between measures of poroviscoelasticity parameters (elasticity, viscosity and porosity) of liver using iMRE and histopathological features graded by ordinal score
Repeatability of elasticity of liver | 1 day During scheduled brain iMRE examination
  Measure of repeatability of elasticity of liver using iMRE
Repeatability of viscosity of liver | 1 day During scheduled brain iMRE examination
  Measure of repeatability of viscosity of liver using iMRE
Repeatability of porosity of liver | 1 day During scheduled brain iMRE examination
  Measure of repeatability of porosity of liver

CONTACTS AND LOCATIONS:
Overall Officials: Van Houten Elijah, Ing., PhD, Principal Investigator — Centre hospitalier de l'Université de Sherbrooke
Locations (2):
- Canada (2):
  - CRCHUM, Montreal, Quebec
  - CRCHUS, Sherbrooke, Quebec